CLINICAL TRIAL: NCT00797472
Title: A Phase II Open Label, Multicenter, Randomized, Parallel Study Comparing the Efficacy of R-mabHD Alone and a Combination of Adriamycin, Bleomycin, Vinblastine and Dacarbazine (ABVD)in Treating Patients With Hodgkin's Disease.
Brief Title: Study Comparing R-mabHD and a Combination of ABVD in Hodgkin's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: American Scitech International (Other)
Collaborators: Eli Lilly and Company (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Dr. R. Grewal, American Scitech International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASI-HDII 1108
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Hodgkin's Disease
Keywords: Hodgkin's Lymphoma; R-mabHD; ABVD treatment; Hodgkin's Disease
MeSH Terms: conditions — Hodgkin Disease | interventions — Doxorubicin; Bleomycin; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I: R-mabHD (Active Comparator): Anti-hodgkin disease agent
  Interventions: Drug: R-mabHD
- Arm II: ABVD (Active Comparator)
  Interventions: Drug: ABVD

INTERVENTIONS:
Drug: R-mabHD — An intravenous infusion containing R-mabHD 375mg/m2 will be administered over a period of 3 to 8 hours every week for eight weeks in a row.
  Arms: Arm I: R-mabHD
Drug: ABVD — A combination of Adriamycin, Bleomycin, Vinblastine and Dacarbazine (ABVD) will be given intravenously over a period of 3 hours every other week for 12 treatments.
  Other Names: Adriamycin, Bleomycin, Vinblastine, Dacarbazine
  Arms: Arm II: ABVD

SUMMARY:
120 subjects with Hodgkin's disease will be randomly divided into two groups: Group I receiving R-mabHD and Group II receiving a combination of Adriamycin,Bleomycin,Vinblastine and Dacarbazine. R-mabHD will be given once a week for eight weeks in a row. The ABVD combination will be given once every other week for 12 treatments. The hypothesis is that intervention with R-mabHD will lead to a quicker remission of Hodgkin's disease than the intervention with a combination of ABVD.

DETAILED DESCRIPTION:
The primary objective is to compare the efficacy of R-mabHD with a combination therapy of Adriamycin, Bleomycin,Vinblastine and Dacarbazine (ABVD) in bringing about remission of Hodgkin's lymphoma and reduction in tumor size.

Primary Study Endpoint: Primary efficacy criterion is percentage of patients achieving a functional score of 1.

Efficacy evaluation is based on assessment of functional score. At the end of six months, a functional assessment of the tumor will be undertaken to record the score as follows:

Score 1: >/= 50% reduction in size of tumor Score 2: < 50% reduction in size of tumor.

Secondary Study Endpoint: Additional secondary endpoint is the average time to achieve 50% reduction in size of tumor.

120 subjects with Hodgkin's Disease will be divided randomly into two groups. 60 subjects (Group I)will receive R-mabHD by intravenous infusion in a dose of 375mg/m2 once a week for eight weeks in a row. The other half (Group II) will receive a combination of intravenous Adriamycin, Bleomycin, Vinblastine and Dacarbazine every other week for 12 treatments. Enrollment period will be three years and subjects from both genders will be accepted. Subjects should be between the ages of 18 and 65. No healthy volunteers will be accepted. Females who are nursing babies or are pregnant will be excluded from the study. Subjects will be evaluated every month for the first six months and then at one year and then at eighteen months after the baseline visit one.

ELIGIBILITY:
Inclusion Criteria:

1. Must sign an informed consent form
2. Must have histologically proven diagnosis of Hodgkin's lymphoma
3. Both genders and age between 18 and 65
4. Must have adequate bone marrow reserve (ANC.1500/mm3, Platelet>50,000/mm3)
5. Must have bidimensionally measureable disease
6. LVEF >50% by echocardiogram
7. Serum creatinine upto one fold
8. Serum bilirubin upto one fold
9. Hepatitis B surface antigen negative
10. Hodgkin's Disease patients who relapse after radiation therapy alone or surgical treatment alone or both,or previously untreated patients with stage II bulky, III and IV.

Exclusion Criteria:

1. HIV positive
2. Pregnant women and women of child bearing age who are not practising adequate contraception
3. Severe pulmonary disease including COPD and asthma
4. Evidence of other malignancy except superficial nonmelanoma skin carcinoma or carcinoma in situ of the cervix
5. Nursing mothers
6. Uncontrolled active infection
7. concurrent prednisone or other systemic steroid therapy
8. Less than 4 weeks since prior radiotherapy
9. Less than 30 days since prior investigational therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
There will be a reduction in the size of the tumor after initiating treatment. | Six months

SECONDARY OUTCOMES:
There will be an improvement in the general condition of the patient and it will be possible to estimate the event free survival rate. | Eighteen months

CONTACTS AND LOCATIONS:
Overall Officials: Ratna Grewal, M.D., Study Chair — American Scitech International; Prem A Nandiwada, M.D., Principal Investigator — Raritan Bay Medical Center
Locations (1):
- Raritan Bay Medical Center, Englishtown, New Jersey, United States